CLINICAL TRIAL: NCT03841032
Title: 4 Week In-Use Study Evaluating the Tolerability of a Skin Care Product on Adults With Rosacea
Brief Title: 4 Week In-Use Study Evaluating How Well-Tolerated a Skin Care Product Is on Adults With Facial Redness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20516
Record Dates: First submitted 2019-01-22; First posted 2019-02-15 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Rosacea
Keywords: Facial redness; Skin sensitivity
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Sunscreen Lotion (Experimental): Subjects with rosacea will apply the test sunscreen lotion to the face for 4 weeks
  Interventions: Drug: Coppertone, BAY1183345

INTERVENTIONS:
Drug: Coppertone, BAY1183345 — Lotion, for 4 weeks

SUMMARY:
The purpose of this study is to evaluate if the test sunscreen skin care product will be well-tolerated and help facial redness when applied to the face after 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or females at least 18 years of age;
* Women of childbearing potential must agree to use adequate contraception when sexually active. Acceptable methods of contraception include, but are not limited to, (i) condoms (male or female) with or without a spermicidal agent; (ii) diaphragm or cervical cap with spermicide; (iii) intra-uterine device; (iv) hormone-based contraception (stable dose for 3 months); (v) partner vasectomy.
* Subjects with general good health as determined by a medical history form;
* Subjects with erythematotelangiectatic and/or papulopustular rosacea, at the baseline evaluation, as determined by the Investigator;
* Subjects with Fitzpatrick Skin Types I through III, as determined by the dermatologist;
* Subjects willing and capable of understanding and providing written informed consent, willing to sign a confidentiality agreement, Health Insurance Portability and Accountability Act (HIPAA) Authorization Form, and to cooperate and participate by following study requirements.

Exclusion Criteria:

* Subjects with only phymatous or ocular rosacea;
* Female subjects of child-bearing potential who test positive in a urine pregnancy test at Baseline (Visit 1), are trying to become pregnant or are nursing;
* Subjects with known allergies to any type of skin care product and/or sunscreen product and/or any ingredients in the test product;
* Subjects with any facial skin disorders which may influence results, in the opinion of the Investigator;
* Subjects with a reported history of acute or chronic dermatological (except for rosacea), uncontrolled hypertension, other medical and/or physical conditions which, in the opinion of the Investigator, interferes with evaluation of the test product or places the subject at risk;
* Subjects currently using medications or oral supplements which, in the opinion of the Investigator, may influence the outcome of the study or interfere with study observations, including rosacea treatment products;
* Individuals using or who have used any systemic medication considered to affect rosacea, specifically, but not exclusively, antibiotics or steroids, who do not agree to continue taking the specified medication at the same dose and regimen throughout the study;
* Subjects who started hormone replacement therapies (HRT) or hormones for birth control less than 3 months prior to study entry or who plan on starting, stopping, or changing doses of HRT or hormones for birth control during the study;
* Subjects with excessive facial hair that would, in the opinion of the Investigator, interfere with diagnosis or assessment of rosacea;
* Subjects who spend excessive time out in the sun;
* Subjects that have received or used an Investigational New Drug within 30 days prior to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Number of subjects exhibiting increases in papules | Up to 4 weeks
Number of subjects exhibiting increases in erythema | Up to 4 weeks
Number of subjects exhibiting increases in dryness, telangiectasia and tactile surface roughness | Up to 4 weeks
Number of subjects exhibiting increases in any subjective irritation | Up to 4 weeks

SECONDARY OUTCOMES:
Change in facial redness measured by spectrophotometer | From baseline up to 4 weeks
Change in facial redness measured by digital imaging | From baseline up to 4 weeks
Percentages for each response to hedonic questionnaire assessing product experience | Up to 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The Education & Research Foundation, Inc., Lynchburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.